CLINICAL TRIAL: NCT07342270
Title: Sensorimotor Psychotherapy for Personality Disorders
Acronym: SPiPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tilburg University (Other)
Collaborators: GGZ Breburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSB_RP2165; NL-009734 (Other: Medisch Ethische Toetsingscommissie Brabant)
Record Dates: First submitted 2025-12-18; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-09

CONDITIONS: Early Chilhood Trauma; Personality Disorder
Keywords: Sensorimotor Psychotherapy; Personality disorders; Early childhood trauma; SP-protocol
MeSH Terms: conditions — Personality Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual for personality disoders
  Interventions: Other: Treatment as ususal
- Sensorimotor Psychotherapy (Experimental): Sensorimotor Psychotherapy 12-session group protocol
  Interventions: Other: Sensorimotor Psychotherapy

INTERVENTIONS:
Other: Sensorimotor Psychotherapy — Sensorimotor psychotherapy (SP) is a body-oriented approach for people with personality disorders. The SP-intervention consists of 12-session SP-protocol which is applied in a groupsetting. Each session starts with psycho-education on a trauma-related topic, followed by one or multiple skills which are practized and discussed within the group.
  Arms: Sensorimotor Psychotherapy
Other: Treatment as ususal — The control condition consists of the standard treatment for personality disorders as provided within the mental health care institution. This treatment may comprise various components, depending on the specific institution. The nature and extent of the treatment provided will be documented.
  Arms: Treatment as usual

SUMMARY:
SUMMARY

Rationale: Personality disorders are treated conform the Dutch GGZ-zorgstandaard mainly with verbal psychotherapies but experts by experience call out to make use of body-oriented approaches as well. In general, the rationale to study the effects of bodily centered therapy for personality disorders is built on the overlap between personality disorders and posttraumatic stress disorder (PTSD). In both classifications, childhood major events and/or traumatic life events play a role in the history of its origins (Karatzias et al., 2023).Traditional psychotherapies for personality disorders address the cognitive and emotional elements of trauma, but lack techniques that work directly with the physiological elements, although trauma profoundly affects the body and many symptoms of traumatized individuals with personality disorders are somatically based. However, studies into the effect of body centered interventions for personality disorders are scarce. This study aims to examine the effects of sensorimotor psychotherapy (SP), a body-oriented intervention, in patients with a personality disorder and PTSD-symptoms. This study studies the effect of sensorimotor psychotherapy (SP) which is a body-oriented intervention which focuses on the combination of a personality disorder and post-traumatic stress disorder.

Objective: This multi-center randomized controlled study aims to research the effect of a 12-session sensorimotor psychotherapy (SP) group intervention, in comparison with treatment-as-usual, on emotion regulation in people with a personality disorder. In addition, the effects on body awareness, self-soothing, PTSD-symptoms and personality functioning are assessed. Patients' perception of the intervention will be assessed through qualitative techniques. The study will be carried out in five mental health institutions in the Netherlands.

Study design: This is a multi-center randomized controlled trial, in which the intervention group receives a 12-sessions SP-therapy, and the control group receives treatment-as-usual of the assigned institution. Measurements through standardized instruments take place at three moments: pre-intervention (T0), post-intervention (T1), and two months follow-up (T2). Qualitative interviews are conducted after completion of the SP-condition. In combination with the qualitative measurements, a Mixed Methods Design is used.

Study population: Patients older than 18 years, who have been diagnosed with a personality disorder and have experienced early childhood trauma.

Intervention: patients assigned to the SP-condition receive the 12-session SP group protocol (Fisher & Ogden, 2016), this protocol introduces diverse successive skills, aiming for the patient to have more somatic resources to regulate arousal of the autonomous nervous system. Every session starts with psychoeducation on a trauma-related theme, followed by one or multiple skills which are practiced in dyads and are later discussed in the group. The subjects which are covered are: autonomous arousal, implicit memory, regulation techniques, survival sources, somatic and internal resources, boundaries, practicing with experiments and repetitions, focus on positive change.

Main study parameter: The main parameter of this study is emotion regulation. Emotion regulation is examined with the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF).

Secondary parameters: Second parameters are body awareness, self-soothing, PTSD-symptoms, personality functioning. Body awareness is examined with the Multidimensional Assessment of Interoceptive Awareness (MAIA-2). The Soothing Receptivity Scale (SRS) is used to examine self-soothing abilities. The PTSD-checklist for DSM-5 (PCL-5) is used to assess the PTSD-symptoms. The Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF 2.0) is used to map out personality functioning. The patients' perception of the intervention is explored through qualitative interviews. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients involved in this study are indicated for treatment for a personality disorder. Sensorimotor psychotherapy belongs the treatment options of some mental health institutions. Additionally, patients who are assigned to the control condition are offered the SP-condition after completing the control condition. In this way they can also benefit from the SP-condition.

Questionnaires are filled in at three moments during the treatment (T0, T1, T2), filling in the questionnaires will take 60 minutes on average, which is little more than routine outcome measurement takes in Dutch mental healthcare. The qualitative interviews after the SP-condition will take up 60 minutes on average.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 and older
* Diagnosed with a personality disorder according to the DSM-classification
* Has a history of early childhood trauma

Exclusion Criteria:

* Does not master Dutch / English sufficiently for filling out the questionnaire cannot fill participate in the research.
* Presents factors or behaviour that disrupts participation in the group and undermines treatment will be excluded from this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotion regulation-Difficulties in Emotion Regulation Scale | A pre-intervention, post-intervention and follow-up (8-weeks post-intervention).
  The Difficulties in Emotion Regulation Scale (DERS) is used to assess the primary parameter, emotion regulation (Kaufman et al., 2016). This is a 36 item self-report questionnaire for evaluating emotion regulation problems. The factors correspond to the six factors from the scale. The scales are: 1. not accepting emotional responses, 2. difficulties in showing goal-directed behavior, 3. problems with impulse control, 4. lack of emotional awareness, 5. limited access to emotion regulation strategies, and 6. lack of emotional clarity. The questionnaire has excellent validity and reliability (Cronbach's alpha = 0.89) (Kaufman et al., 2016). A higher score indicates more problems in emotion regulation.

SECONDARY OUTCOMES:
Body awareness- Multidimensional Assessment of Interoceptive Awareness | A pre-intervention, post-intervention and follow-up (8-weeks post-intervention).
  Multidimensional Assessment of Interoceptive Awareness (MAIA-2) (Mehling et al., 2018) is used to assess the extent of body awareness. This is a 37-item self-report questionnaire with a 6-point Likert scale focusing on interoceptive awareness. There are 8 subscales: noticing, not-distracting, not-overthinking, attention regulation, emotional awareness, self-regulation, body awareness and confidence. Cronbach's alpha varies from 0.67 to 0.89 on the subscales and factor structure is confirmed (Mehling et al., 2015; Scheffers et al., 2024). A higher score indicates more body awareness.
Self-soothing-Soothing Receptivity Scale | A pre-intervention, post-intervention and follow-up (8-weeks post-intervention).
  Soothing Receptivity Scale (SRS) (Glassman, 1988) is used to assess receptivity to calm. This is a 27-item self-report questionnaire with a 5-point Likert scale to assess the experience being calmed down, being physically calmed down, the experience of calming down by sharing emotions with others and self-soothing. The SRS has good internal consistency (Cronbach's alpha = 0,80). The higher the score, the more capable one is to self-sooth.
PTSD-symptoms - PTSD-checklist for DSM-5 | A pre-intervention, post-intervention and follow-up (8-weeks post-intervention).
  PTSD-checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire which questions symptoms of PTSD on a 5-point Likert Scale with a good reliability (Cronbach's alpha =0.94), test-retest reliability and discriminating validity (Blevins et al., 2015). A change of 5 points is seen as a relevant change during treatment. A change of 10 points in total score is a minimum for clinical relevant changes.
Level of Personality functioning - Level of Personality Functioning Scale-Brief Form 2.0 | A pre-intervention, post-intervention and follow-up (8-weeks post-intervention).
  Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF 2.0) (Weekers et al.,2019) assesses personality functioning. The LPFS-BF is a 12-item self-report questionnaire with a 4-point Likert Scale and gives the general severity of the personality pathology based on the Alternative Model for Personality disorder from section III of the DSM-5. The items are clustered in two higher domains, Self-functioning and Interpersonal functioning. The questionnaire is sufficient reliability and is sensitive for change. A score higher than 2 on one of the two domains refers to problems in personality functioning. A higher score indicates more disfunctioning.